CLINICAL TRIAL: NCT01991652
Title: Collaborative Wilms Tumour Africa Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Trijn Israels, Paediatric Oncologist, MD PhD, Amsterdam UMC, location VUmc
Other Study IDs: CollabWilmsAfrica
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Wilms Tumour
Keywords: Wilms tumour; Childhood cancer; Africa
MeSH Terms: conditions — Wilms Tumor; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Wilms tumour: Children diagnosed with a Wilms tumour receive SIOP PODC Wilms tumour treatment; preoperative chemotherapy, surgery and postoperative chemotherapy (= standard care).
  One group of patients.

SUMMARY:
Significant progress has been made in the treatment of Wilms tumor in high income countries, where survival is now around 85% - 90%. Survival in low income countries is much lower; specific challenges include late presentation, malnutrition, less intense supportive care facilities and failure to complete treatment.

A comprehensive treatment guideline was introduced in Malawi in 2006 which included nutritional support and social support to enable parents to complete treatment. Survival has increased to around 50%; 95% of children completed their treatment. A multi-disciplinary group of African clinicians and 'state of the art' experts produced a consensus treatment guideline for children with Wilms tumor in sub-Saharan Africa. This guideline will be implemented as a multi-center prospective clinical trial in 2014 in six - eight institutes, expecting about 200 new patients per year.

The hypothesis is that 2 year event free survival will be 50%, with <10% failure to complete treatment and <10% treatment related mortality. Other research questions include efficacy and toxicity of preoperative chemotherapy and the comparison of surgical staging, local pathology and central review pathology in stratifying postoperative chemotherapy.

DETAILED DESCRIPTION:
Patients are treated according to standard care. Data are documented on presentation at diagnosis, response of the tumor, findings at surgery and pathology, treatment given and outcome of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years
* Diagnosis Wilms tumour

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children (< 18 years) diagnosed with a Willms tumour
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 2 years
  Percentage of patients with no event after two years of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Trijn Israels, MD PhD, Study Chair — Amsterdam UMC, location VUmc
Locations (3):
- Mbingo Mission Hospital, Bamenda, Cameroon
- Korle Bu Hospital, Accra, Ghana
- College of Medicine, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Israels T, Moreira C, Scanlan T, Molyneux L, Kampondeni S, Hesseling P, Heij H, Borgstein E, Vujanic G, Pritchard-Jones K, Hadley L. SIOP PODC: clinical guidelines for the management of children with Wilms tumour in a low income setting. Pediatr Blood Cancer. 2013 Jan;60(1):5-11. doi: 10.1002/pbc.24321. Epub 2012 Sep 26. PMID 23015404
- [Result] Israels T, Renner L, Hendricks M, Hesseling P, Howard S, Molyneux E; Paediatric Oncology in Developing Countries. SIOP PODC: recommendations for supportive care of children with cancer in a low-income setting. Pediatr Blood Cancer. 2013 Jun;60(6):899-904. doi: 10.1002/pbc.24501. Epub 2013 Feb 25. PMID 23441092
- [Result] Israels T, Kambugu J, Kouya F, El-Mallawany NK, Hesseling PB, Kaspers GJ, Eden T, Renner L, Molyneux EM. Clinical trials to improve childhood cancer care and survival in sub-Saharan Africa. Nat Rev Clin Oncol. 2013 Oct;10(10):599-604. doi: 10.1038/nrclinonc.2013.137. Epub 2013 Jul 30. PMID 23897077